CLINICAL TRIAL: NCT03431805
Title: TRAnexamic Acid for Preventing Postpartum Hemorrhage Following a Cesarean Delivery :a Multicenter Randomised, Double Blind Placebo Controlled Trial (TRAAP2)
Brief Title: TRAnexamic Acid for Preventing Postpartum Hemorrhage Following a Cesarean Delivery
Acronym: TRAAP2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CHUBX 2015/41
Record Dates: First submitted 2018-01-30; First posted 2018-02-13 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Postpartum Hemorrhage
Keywords: Randomized; double blind placebo controlled trial; prevention; tranexamic acid; postpartum hemorrhage; cesarean
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid (Experimental): intravenous administration of 10-mL of tranexamic acid (EXACYL® 1 g/10 ml I.V., solution injectable)
  Interventions: Drug: Tranexamic Acid Injectable Solution
- Chloride solution (Placebo Comparator): sodium intravenous administration of 10-mL of chloride solution (0.9% -10mL).
  Interventions: Drug: Sodium Chloride 0.9%

INTERVENTIONS:
Drug: Tranexamic Acid Injectable Solution — After the routine and prophylactic administration of a uterotonic , the intervention will be the IV administration of a 10-ml blinded ampoule of the study drug (either TXA or placebo according to the randomisation sequence) to the woman within 3 minutes after birth, slowly (over 30-60 seconds), once the cord has been clamped.
  Arms: Tranexamic acid
Drug: Sodium Chloride 0.9% — After a routine and prophylactic administration of a uterotonic , the intervention will be the IV administration of a 10-ml blinded ampoule of the study drug (either TXA or placebo according to the randomisation sequence) to the patient within 3 minutes afterbirth), slowly (over 30-60 seconds), once the cord has been clamped.
  Arms: Chloride solution

SUMMARY:
The aim is to assess the impact of tranexamic acid (TXA) for preventing postpartum hemorrhage (PPH) following a cesarean section (CS).

DETAILED DESCRIPTION:
Regarding the prevention of PPH, recent randomized controlled trials (RCTs) of unclear quality have suggested that TXA may reduce blood loss and maternal morbidity, while a Cochrane Collaboration review has concluded, that "TXA (in addition to uterotonic medications) decreases postpartum blood loss and prevents PPH and blood transfusions following vaginal birth and CS in women at low risk of PPH based on studies of mixed quality. Further investigations are needed on efficacy and safety of this regimen for preventing PPH.

Treatment, that is a 10-mL blinded vial of the study drug (either 1g TXA or placebo according to the randomization sequence), will be administered intravenously to the participant women during the third stage of labor of cesarean delivery.

The follow-up visit will take place in the postpartum ward of the maternity unit, on D2 postpartum. This stage will include a venous blood sample to measure plasma concentrations of Hb and Ht, urea and creatinemia, prothrombin time (PT), active prothrombin time (aPTT), aspartate and alanine transaminase, total bilirubin and fibrinogen, and the completion of a self-questionnaire about satisfaction by the women, as well as the assessment of the adverse events.

At 8 weeks postpartum, a self-questionnaire assessing psychological status and well-being will be sent to the women. At 12 weeks postpartum, all participants will be contacted by phone to assess the incidence of thrombotic and any other significant events.

ELIGIBILITY:
Inclusion Criteria:

* : adult women admitted for a cesarean delivery before or during labor, at a term ≥ 34 weeks,
* hemoglobin level at the last blood sample >9g/dl,
* available blood test for Hb and Ht within one week before caesarean delivery,
* informed signed consent

Exclusion Criteria:

* previous thrombotic event or preexisting pro-thrombotic disease,
* epileptic state or history of seizures,
* presence of any chronic or active cardiovascular disease outside hypertension,
* any chronic or active renal disease and chronic or active liver disease at risk thrombotic or hemorrhagic, autoimmune disease,
* sickle cell disease,
* placenta praevia,
* placenta accreta/increta/percreta,
* abruption placentae,
* eclampsia,
* HELLP syndrome,
* significant hemorrhage before cesarean section
* in utero fetal death,
* administration of low-molecular-weight heparin or antiplatelet agents during the week before delivery,
* planned general anesthesia,
* hypersensitivity to tranexamic acid or concentrated hydrochloric acid,
* instrumental extraction failure,
* multiple pregnancy with vaginal delivery of the first child,
* poor understanding of the French language.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4574 (Actual)
Dates: Start 2018-03-03 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
postpartum hemorrhage | day 2
  Incidence of PPH defined by a calculated blood loss > 1000mL [Calculated estimated blood loss = estimated blood volume × (preoperative Ht - postoperative Ht)/preoperative Ht (where estimated blood volume (mL) = weight (Kg) × 85)] or red blood cell transfusion up to day 2 postpartum. Preoperative Ht will be the most recent Ht within one week before delivery. Postoperative Ht will be measured at D2

SECONDARY OUTCOMES:
mean calculated blood loss > 500mL | day 2
mean calculated blood loss > 1500mL | day 2
total mean calculated blood loss | day 2
mean gravimetrically estimated blood loss | 6 hours
  by measuring the suction volume and swab weight; proportion of women requiring supplementary uterotonic treatment including sulprostone
incidence of postpartum transfusion | day 2
Mean or median number of units of red blood cells transfused | day 2
incidence of arterial embolisation or emergency surgery for PPH | 3 months
mean peripartum change in haemoglobin | day 2
  difference between the most recent Hb within one week before delivery and at day 2 postpartum
mean peripartum change in hematocrit | day 2
  difference between the most recent Ht within one week before delivery and at day 2 postpartum
heart rate | 15, 30, 45, 60 and 120 minutes after delivery
  bpm
diastolic blood pressure | 15, 30, 45, 60 and 120 minutes after delivery
  mmHg
systolic blood pressure | 15, 30, 45, 60 and 120 minutes after delivery
  mmHg
number of participants with nausea reported by caregivers | 6 hours
number of participants with vomiting reported by caregivers | 6 hours
number of participants with phosphenes reported by caregivers | 6 hours
number of participants with dizziness reported by caregivers | 6 hours
creatinemia | day 2
  micromol/L
urea | day 2
  g/L
prothrombin time (PT) | day 2
aspartate transaminase | day 2
  IU/L
alanine transaminase | day 2
  IU/L
total bilirubin | day 2
  micromol/L
total fibrinogen | day 2
  g/L
number of participants with deep venous thrombosis confirmed by paraclinical exams | within twelve weeks after the delivery
number of participants with pulmonary embolism confirmed by paraclinical exams | within twelve weeks after the delivery
number of participants with myocardial infarction confirmed by paraclinical exams | within twelve weeks after the delivery
number of participants with any thrombotic event confirmed by paraclinical exams | within twelve weeks after the delivery
seizure | within twelve weeks after the delivery
renal failure | within twelve weeks after the delivery
  defined by the need for dialysis
women's satisfaction | day 2 and weeks 8 postpartum
  assessed by a self-administered questionnaire
Provider-assessed clinically significant PPH | day 2
Hb drop > 2g/DL | day 2
Active prothrombin time (aPTT) | day 2
aspartate transaminase > 2N | day 2
alanine transaminase > 2N (day 2) | day 2
gravimetrically estimated blood loss > 500mL | day 2
gravimetrically estimated blood loss > 1000 mL | day 2
Shock | day 2
Transfer to Intensive Care Unit | twelve weeks after delivery
Death from any cause | 42 days postpartum
supplementary uterotonic treatment | day 2
  proportion of women requiring supplementary uterotonic treatment
iron sucrose perfusion | discharge from hospital
  incidence of iron sucrose perfusion
mean gravimetrically estimated blood loss | at the end of the cesarean delivery

CONTACTS AND LOCATIONS:
Locations (26):
- France (26):
  - CHU Angers, Angers
  - CHU Jean Minjoz, Besançon
  - CHU Bordeaux, Bordeaux
  - CHRU Côte de Nacre, Caen
  - CHU Estain, Clermont-Ferrand
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Hôpital Saint Joseph Marseille, Marseille
  - Hopital Nord, Marseille
  - CHU de Montpellier, Montpellier
  - CHRU de Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Nîmes, Nîmes
  - Hôpital Trousseau, Paris
  - Hôpital Saint Joseph Paris, Paris
  - Maternité de Port-Royal Paris, Paris
  - Hôpital universitaire Necker-Enfants malades, Paris
  - Hôpital universitaire Robert Debré, Paris
  - Hôpital universitaire Kremlin-Bicètre, Paris
  - CH de Pau, Pau
  - Centre Hospitalier Intercommunal Poissy-Saint Germain, Poissy
  - CHU Rennes, Rennes
  - CHU Charles Nicolle, Rouen
  - CHU Saint Etienne, Saint-Etienne
  - CHU Strasbourg, Strasbourg
  - Hôpital Paule de Viguier CHU Toulouse, Toulouse
  - CHU Tours, Tours

REFERENCES:
- [Derived] Sentilhes L, Benard A, Madar H, Froeliger A, Petit S, Deneux-Tharaux C; TRAAP2 study group. Tranexamic acid for reduction of blood loss after Caesarean delivery: a cost-effectiveness analysis of the TRAAP2 trial. Br J Anaesth. 2023 Nov;131(5):893-900. doi: 10.1016/j.bja.2023.07.028. Epub 2023 Sep 9. PMID 37690946
- [Derived] Sentilhes L, Senat MV, Le Lous M, Winer N, Rozenberg P, Kayem G, Verspyck E, Fuchs F, Azria E, Gallot D, Korb D, Desbriere R, Le Ray C, Chauleur C, de Marcillac F, Perrotin F, Parant O, Salomon LJ, Gauchotte E, Bretelle F, Sananes N, Bohec C, Mottet N, Legendre G, Letouzey V, Haddad B, Vardon D, Madar H, Mattuizzi A, Daniel V, Regueme S, Roussillon C, Benard A, Georget A, Darsonval A, Deneux-Tharaux C; Groupe de Recherche en Obstetrique et Gynecologie. Tranexamic Acid for the Prevention of Blood Loss after Cesarean Delivery. N Engl J Med. 2021 Apr 29;384(17):1623-1634. doi: 10.1056/NEJMoa2028788. PMID 33913639
- [Derived] Sentilhes L, Daniel V, Deneux-Tharaux C; TRAAP2 Study Group and the Groupe de Recherche en Obstetrique et Gynecologie (GROG). TRAAP2 - TRAnexamic Acid for Preventing postpartum hemorrhage after cesarean delivery: a multicenter randomized, doubleblind, placebo- controlled trial - a study protocol. BMC Pregnancy Childbirth. 2020 Jan 31;20(1):63. doi: 10.1186/s12884-019-2718-4. PMID 32005192